CLINICAL TRIAL: NCT02058849
Title: Randomized Phase II Study of Concentrated Beet Root in Participants Being Treated for Locally Advanced Unresectable, Previously Untreated Squamous Cell Cancer of the Head and Neck
Brief Title: Randomized Study of Beet Root in Locally Advanced Squamous Cell Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Travis Thomas (Other)
Responsible Party: Sponsor-Investigator, David Travis Thomas, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-HN-23-MCC
Record Dates: First submitted 2014-01-23; First posted 2014-02-10 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Mucositis
Keywords: Mucositis; Beetroot; Head and neck cancer
MeSH Terms: conditions — Mucositis; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Beetroot (Experimental): Beetroot 10 grams concentrated organic beetroot crystals
  Interventions: Drug: Beetroot
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Beetroot — 10g Beetroot powder mixed with 4-8 oz.
  Other Names: BEETELITE™ NeO Shot
  Arms: Beetroot
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of the current proposal is to determine if concentrated beet root could improve medical treatment compliance as defined by completion of radiotherapy and 3 cycles of chemoradiation without dose reduction, preserve fat-free mass, and strength while reducing mucositis. The investigators central hypothesis is that dietary nitrate supplementation in head and neck cancer patients receiving aggressive medical care will improve compliance with medical treatment by attenuating the loss of muscle mass and strength and reducing symptoms (mucositis) associated with treatment compared to patients receiving standard care with placebo.

DETAILED DESCRIPTION:
This is a parallel 2-arm, 1:1 pilot randomized, placebo controlled supplementation study designed to examine improvements in chemoradiation compliance, body composition, strength/endurance, quality of life, nutrition status, and mucositis symptoms by supplementing beetroot juice over a period of 12 weeks. The Investigators plan to recruit 50 individuals with squamous cell carcinoma of the head and neck who are planning to undergo chemoradiation/intensity-modulated radiation therapy (IMRT). All subjects will be over 18 years of age. Eastern Cooperative Oncology Group (ECOG) performance status should be less than or equal to 2, which is necessary to ensure the patient can adequately participate in the supplementation and planned test procedures. All eligible participants will have a life expectancy greater than or equal to 3 months and normal organ and marrow function at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically squamous cell carcinoma of the head and neck and be planned for definitive radiation and chemotherapy.
* Patients must have not received prior radiotherapy or chemotherapy for the current head and neck cancer. Patients may have a history of prior malignancy, but must be able to tolerate full dose radiation and chemotherapy for the current head and neck cancer, as determined by the treating oncologist.
* Age ≥18 years.
* ECOG performance status ≤2
* Life expectancy of greater than 3 months
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ 1.5 times ULN (upper limit of normal)
  * ALT and AST ≤ 2.5 times the ULN
  * Creatinine ≤ 1.5 times ULN OR
  * Measured creatinine clearance > 60 mL/min
  * Able to swallow thin liquids or have a feeding tube for delivery of nutrition.
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active serious infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled cardiac arrhythmia
  * Uncontrolled hypertension
  * Psychiatric illness or social situation that would preclude compliance with study
* No other concurrent investigational or anticancer therapies or agents.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of beet root administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Active infection > CTCAE Grade 2, that is considered clinically serious by the treating physician.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study dietary supplement.
* Patients who are receiving any other investigational agents.
* Pregnant women are excluded from this study because chemo-radiation has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemoradiation, breastfeeding should be discontinued.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with beet root.
* Subjects with a history of calcium oxalate nephrolithiasis.
* Subjects with a significant history of malabsorption (e.g. celiac sprue, short bowel syndrome, or other, as determined by the treating physician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis Thomas, PH.D., RD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Beetroot | Placebo
Started | 11 | 2
Completed | 4 | 1
Not Completed | 7 | 1
Not completed — Hospitalization | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beetroot | Placebo | Total
Number analyzed (Participants) | 11 | 2 | 13
Age, Continuous [Median (Full Range); unit: years] | 53 [45 to 67] | 49 [47 to 51] | 51 [45 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 9 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 2 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Treatment
Description: Number of patients completing radiotherapy and three cycles of chemotherapy with no delay
Time Frame: Up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 4 | 1

2. Primary Outcome: Endurance
Description: Biodex endurance peak torque (Nm)
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
Nm
  Baseline (1-2 weeks pre-IMRT) | 161.2 (31.3) | 129
  Midpoint (7-8 weeks following IMRT initiation) | 116.0 (22.2) | 139.8
  Endpoint (4-6 weeks following Midpoint) | 122.7 (23.5) | 95.2

3. Secondary Outcome: Body Composition (Lean Body Mass)
Description: Grams of lean body mass
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
grams
  Baseline (1-2 weeks pre-IMRT) | 59245.3 (11120.8) | 63469
  Midpoint (7-8 weeks following IMRT initiation) | 51524.0 (10650.5) | 60833
  Endpoint (4-6 weeks following Midpoint) | 52170.0 (10969.9) | 57005

4. Secondary Outcome: Muscle Strength
Description: Peak force (Nm) from one-legged maximum voluntary contraction (MVC) using the Biodex isokinetic machine.
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Population: Midpoint data were not collected from the placebo group for this outcome.
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
Nm
  Baseline (1-2 weeks pre-IMRT) | 176.1 (4.2) | 120.3
  Midpoint (7-8 weeks following IMRT initiation) | 149.8 (26.1) | NA — Midpoint data were not collected from the placebo group for this outcome.
  Endpoint (4-6 weeks following Midpoint) | 162.6 (27.5) | 133.6

5. Other Pre Specified Outcome: Handgrip Strength
Description: Peak force (kg) measured using a handgrip dynamometer
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
kg
  Baseline (1-2 weeks pre-IMRT) | 53.2 (12.3) | 35
  Midpoint (7-8 weeks following IMRT initiation) | 48.2 (12.0) | 33.3
  Endpoint (4-6 weeks following Midpoint) | 46.8 (10.9) | 32.5

6. Other Pre Specified Outcome: Handgrip Strength at 30 Seconds
Description: Handgrip strength (kg) at 30 seconds measured using a handgrip dynamometer
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
kg
  Baseline (1-2 weeks pre-IMRT) | 28.7 (2.7) | 18
  Midpoint (7-8 weeks following IMRT initiation) | 26.7 (3.6) | 21.5
  Endpoint (4-6 weeks following Midpoint) | 25.0 (9.7) | 22.5

7. Other Pre Specified Outcome: Body Fat
Description: Grams of body fat
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
grams
  Baseline (1-2 weeks pre-IMRT) | 29478.8 (11003.8) | 44528
  Midpoint (7-8 weeks following IMRT initiation) | 27093.3 (10889.1) | 45419
  Endpoint (4-6 weeks following Midpoint) | 26075.5 (9173.5) | 37713

8. Other Pre Specified Outcome: Bone Mineral Content
Description: Bone mineral content (grams).
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
grams
  Baseline (1-2 weeks pre-IMRT) | 3011.7 (569.7) | 3728
  Midpoint (7-8 weeks following IMRT initiation) | 2651.5 (664.4) | 3719
  Endpoint (4-6 weeks following Midpoint) | 2020.5 (1315.7) | 3668

9. Other Pre Specified Outcome: Bone Mineral Density
Description: Bone mineral density (grams per centimeter squared)
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Population: Midpoint data were not collected from the placebo group for this outcome.
Measure: Mean (Standard Deviation); unit: grams per centimeter squared
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
grams per centimeter squared
  Baseline (1-2 weeks pre-IMRT) | 1.2 (0.2) | 1.4
  Midpoint (7-8 weeks following IMRT initiation) | 1.1 (0.2) | NA — Midpoint data were not collected from the placebo group for this outcome.
  Endpoint (4-6 weeks following Midpoint) | 1.1 (0.2) | 1.3

10. Other Pre Specified Outcome: Fat Free Mass
Description: Kilograms of fat free mass
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Population: Midpoint data were not collected from the placebo group for this outcome.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
kilograms
  Baseline (1-2 weeks pre-IMRT) | 28.1 (9.4) | 67.2
  Midpoint (7-8 weeks following IMRT initiation) | 27.7 (11.9) | NA — Midpoint data were not collected from the placebo group for this outcome.
  Endpoint (4-6 weeks following Midpoint) | 35.8 (22.1) | 37.7

11. Other Pre Specified Outcome: Total Body Mass
Description: Kilograms of body mass
Time Frame: Baseline (1-2 weeks pre-IMRT), Midpoint (7-8 weeks following IMRT initiation), Endpoint (4-6 weeks following Midpoint).
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Beetroot | Placebo
Number analyzed (Participants) | 4 | 1
kilograms
  Baseline (1-2 weeks pre-IMRT) | 87.4 (19.9) | 111.7
  Midpoint (7-8 weeks following IMRT initiation) | 81.3 (14.7) | NA — Midpoint data were not collected from the placebo group for this outcome.
  Endpoint (4-6 weeks following Midpoint) | 80.9 (12.8) | 98.4

ADVERSE EVENTS:
Time Frame: 4 months
Description: see protocol
Arm/Group | Beetroot | Placebo
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/2
Other Adverse Events (participants affected / at risk) | 9/11 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beetroot (N=11) | Placebo (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 9 (10) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 0 (0)
Oral pain (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (6) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial ended with only one participant in the placebo group. Intra-group and comparative statistics were thus not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02058849/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02058849/ICF_001.pdf